CLINICAL TRIAL: NCT04205578
Title: A Multi-center, Randomized, Single-blind, Placebo-controlled Study of Dl-3-n-butylphthalide in Patients With Moyamoya Disease of High Risk for Ischemic Cerebrovascular Events After Extracranial-to-intracranial Revascularization Surgery
Brief Title: NBP in Patients With Moyamoya Disease of High Risk for Ischemic Cerebrovascular Events
Acronym: NICE-MMD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: yuanli Zhao (Other)
Collaborators: Peking University International Hospital (Other)
Responsible Party: Sponsor-Investigator, yuanli Zhao, Professor, Department of Neurosurgery, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KY2019-023
Record Dates: First submitted 2019-12-18; First posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Moyamoya Disease; Ischemic Cerebral Infarction; Ischemic Stroke; Ischemic Cerebrovascular Accident; Transient Ischemic Attack
Keywords: Dl-3-n-butylphthalide; Revascularization surgery; Extracranial-to-intracranial revascularization; Direct bypass surgery; Combined bypass surgery; Indirect bypass surgery
MeSH Terms: conditions — Moyamoya Disease; Ischemic Stroke; Ischemic Attack, Transient | interventions — 3-n-butylphthalide; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Butylphthalide (NBP) (Active Comparator): For patients without obvious intracranial hemorrhage on CT scan at 4 hours after surgery, 25 mg of NBP in 100 mL of normal saline was administered intravenously since the day of surgery and continued twice daily for 14 postoperative days.
  Interventions: Drug: dl-3-n-butylphthalide (NBP)
- Normal saline (Placebo Comparator): For patients without obvious intracranial hemorrhage on CT scan at 4 hours after surgery, 100 mL of normal saline was administered intravenously since the day of surgery and continued twice daily for 14 postoperative days.
  Interventions: Drug: Normal Saline 0.9% Infusion Solution

INTERVENTIONS:
Drug: dl-3-n-butylphthalide (NBP) — 25 mg of NBP in 100 mL of normal saline was administered intravenously since the day of extracranial-to-intracranial bypass surgery and continued twice daily for 14 postoperative days.
  Arms: Butylphthalide (NBP)
Drug: Normal Saline 0.9% Infusion Solution — 100 mL of normal saline was administered intravenously since the day of extracranial-to-intracranial bypass surgery and continued twice daily for 14 postoperative days.
  Arms: Normal saline

SUMMARY:
An extracranial-to-intracranial (EC-IC) revascularization is the most widely used treatment to improve cerebral perfusion in patients with moyamoya disease (MMD), and it has been shown to reduce the risk of subsequent stroke and neurological deficit. However, perioperative changes in cerebral hemodynamics can induce fluctuations in cerebral perfusion that may lead to transient or irreversible neurological deficits. Our preliminary single-center study suggests that postoperative intravenous administration of dl-3-n-butylphthalide (NBP) may alleviate perioperative neurological deficits and improve the neurological outcomes after EC-IC revascularization for MMD. This is a multicenter, randomized, double-blind, single-controlled, add-on to standard of care study of NBP in patients with MMD of high risk for ischemic cerebrovascular events after EC-IC revascularization surgery.

DETAILED DESCRIPTION:
This trial is a prospective, randomized, singe-blinded, placebo parallel controlled, multiple-center trial.

A total of approximately 450 patients (age between18 years and 60 years) with moyamoya disease after EC-IC revascularization will be enrolled. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 into two groups after offering informed content: 1) one group will receive butylphthalide in 100 mL of normal saline twice daily since the day of surgery and continued for 14 postoperative days; 2) the other group will receive 100 mL of normal saline twice daily since the day of surgery and continued for 14 postoperative days.

The primary objective is to evaluate the rate and severity of ischemic cerebral event in MMD patients with butylphthalide after EC-IC bypass surgery. The study consists of four visits including the day of randomization(baseline), postoperative day 1 before the first injection, 14 days after surgery when the injection therapy is done, and 30 after suryery. Demographic information, symptoms and signs, laboratory test, neuro-imaging assessment, neurological function scale will be recorded during the program. The rate of stroke event, neurological deficit and severity of neurological deficits will be assessed by modified Rankin scale. The trial is anticipated to last from January 2020 to December 2022 with subjects recruited form two neurosurgical centers in Beijing, China.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 and ≤ 60 years.
2. Women of childbearing potential (WOCBP) must have a negative urine HCG pregnancy test at Screening and be practicing a medically acceptable method of contraception with an annual failure rate of less than 1% until the completion of the trial or 60 days after discontinuation of study treatment. Women are considered not childbearing if they are > 1 year postmenopausal or surgically sterile (ie, hysterectomy, bilateral oophorectomy, or bilateral salpingectomy tubal ligation). If serum bHCG is the standard of care, then this value can be used to determine eligibility.
3. A clinical diagnosis of moyamoya disease, including unilateral and bilateral disease.
4. Previous clinical diagnosis of stroke or transient ischemic attack or undiagnosed infarction evidenced on screening CT or MRI
5. Patients with moyamoya disease underwent extra cranial-to-intracranial (EC-IC) bypass surgery, including direct or indirect or combined EC-IC bypass surgery
6. Capable of understanding the purpose and risk of the study and has signed, in writing, the ICF. If the subject is not capable of this at the time of enrollment, a legally authorized representative will provide written informed consent in accordance with all regulations.
7. Ability to comply with study follow-up.

Exclusion Criteria:

1. Female subjects who are pregnant, lactating/breast-feeding, or plan to become pregnant within the next 3 months.
2. severely disabled, as defined by a Modified Rankin Scale (mRS) score more than 3.
3. History of intracranial hemorrhage.
4. Postoperative intracranial hemorrhage on CT scan at 4 hours after surgery.
5. Dementia or other progressive neurological disease.
6. Known life expectancy < 6 months (for any reason).
7. Known allergy or hypersensitivity to celery.
8. Received treatment with any other investigational drug within 30 days before baseline, was previously treated with NBP, is currently taking celery seed extract, or is currently participating in another clinical study.
9. Persons unable or unlikely to return for follow-up visits.
10. Any other reasons that, in the opinion of the investigator, make the subject unsuitable for enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative ischemic stroke rate | within 30 days after surgery
  Perioperative cerebral stroke was defined as a symptomatic event of new cerebral infarction within 30 days after surgery and confirmed by CT or MRI. Symptoms included focal neurological deficit or headache lasting more than 24 hours.
Perioperative death rate | within 30 days after surgery
  Rate of perioperative death of any cause within 30 days after surgery
Rate of transient neurological deficit (TND) | within 30 days after surgery
  TND was defined as either any reversible neurological deficits observed objectively (e.g., hemiparesis, dysarthria) or any reversible neurological deficits recognized and reported subjectively (e.g., facial palsy), and without evidence of intracranial hemorrhage and cerebral infarction on images

SECONDARY OUTCOMES:
modified Rankin Scale scores at 30 days after surgery | at 30 days after surgery
  The modified Rankin Scale scores were recorded at 1 month after surgery.
The severity of transient neurological deficit | within 30 days after surgery
  The severity of TND was further categorized into four grades based on the clinical symptoms and duration6: Grade 0, none TND; Grade 1, symptoms resolved within 5 days; Grade 2, symptoms prolonged for 5 to 9 days; Grade 3; symptoms prolonged for 10 or more days. One grade worse was scored if there were hemiparesis and/or seizure.
Postoperative intracranial hemorrhagic event | within 30 days after surgery
  New-onset intracranial hemorrhage within 30 days after surgery and confirmed by CT or MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanli Zhao, MD, Study Director — Beijing Tiantan Hospital
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol to be published in peer-reviewed journal
Supporting Information: Study Protocol
Time Frame: Since the publication of study protocol
Access Criteria: Available from the principle investigator upon reasonable request